CLINICAL TRIAL: NCT05795998
Title: Turkish Adaptation of Romantic Relationship Sabotage Scale (T-RSS): Validity and Reliability Study
Brief Title: Turkish Adaptation of Romantic Relationship Sabotage Scale Validity and Reliability Study
Acronym: T-RSS
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Ozgur Maden, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: SultanAbdulhamid Khan RTH
Record Dates: First submitted 2023-02-17; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Unrecognized Condition
Keywords: reliability; romantic relationship; sabotage; scale; validity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adaptation of the Sabotage in Romantic Relationships Scale into Turkish and its validity and reliability analyzes — Approval was obtained from the local ethics committee before starting the study. Permission was obtained from Racquel PEEL, who developed the scale. The scale was administered to 495 participants and they were informed about the study by a specialist psychiatrist. Language validity, construct validity and reliability analyzes of the scale were performed. The findings were discussed in the light of the literature.

SUMMARY:
In this cross-sectional and relationship-seeking study, it was aimed to adapt the Romantic Relationship Sabotage Scale (T-RSS), developed by Racquel Peel, into Turkish, for the reasons why partners sabotage the relationship in romantic relationships.

DETAILED DESCRIPTION:
Semi-structured sociodemographic data form, Sabotage in Romantic Relations Questionnaire (RISA), Self-Sabotage Questionnaire, was given to the participants after the interview to be conducted by volunteers aged 18 and over and having a romantic relationship and a psychiatrist working at the Sultan Abdulhamid Han Training and Research Hospital Mental Health and Diseases Service. The Perceived Romantic Relationship Quality Scale (SRS), the Perceived Romantic Relationship Quality Scale (ARIÖ), and the Attitudes Related to Love Scale (AİTÖ) will be given and they will be asked to fill in these forms. Participants will be divided into three study groups. The first study group will consist of at least 30 people for the Linguistic Equivalence Review of the scale. The second study group will consist of at least 30 people for the Confirmatory Factor Analysis, Equivalent Scale Validity and Cronbach Alpha Internal Consistency Reliability Coefficient Examination of the scale. The third study group will consist of at least 30 people for Test/Retest Reliability Analysis, and the same tests will be re-administered to the participants three weeks later. The selection of the sample will be made by simple random sampling method. The criteria given by Tabachnick and Fidell (2007) for factor analysis will be taken into account in determining the number of the research sample. According to these researchers, 300 people are evaluated as "good", 500 people as "very good" and 1000 people as "excellent" for factor analysis.

Back translation method will be used in the translation study of the Sabotage in Romantic Relations Questionnaire (RISA) (Brislin, 1970). First of all, the original form of the scale will be translated into Turkish by at least three experts with a doctorate degree in psychiatry and/or clinical psychology and at least three English language experts, independently of each other with a good level of English. The created form will be translated back into English by the researchers, a psychiatrist or clinical psychologist and two English Language experts. Both English and Turkish translations of the scale will be brought together by creating a "Language Validity Examination Form" (Seçer, 2015, p. 70) by the researchers. The Language Validity Examination Form will be compared by experts and evaluated in terms of translation suitability, and the final form of the scale will be decided by choosing the most appropriate items that reflect the theoretical structure better and are more linguistically understandable by majority vote.

Analysis of study data will be done using SPSS for Windows 22.0 and AMOS 24.0 package programs. In statistical interpretations, p<.05 values will be considered significant at the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study,
2. Having 18 years or older,
3. Having a romantic relationship
4. Having no problem in reading and understanding the semi-structured socio-demographic data form, the Romantic Relationships Sabotage Scale (RSS), the Self-handicapping Scale (SHS), the Perceived Romantic Relationship Quality Scale (PRRQS), and the Love Attitudes Scale-Short Form (LAS-SF)

Exclusion Criteria:

1. Those who did not volunteer to participate in the study,
2. Having under the age of 18,
3. Those who are not in a romantic relationship D. Those with psychiatric disorders who cannot read and fill in the semi-structured sociodemographic data form, the Romantic Relationships Sabotage Scale (RSS), the Self-handicapping Scale (SHS), the Perceived Romantic Relationship Quality Scale (PRRQS), and the Love Attitudes Scale-Short Form (LAS-SF)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female volunteer participants who applied to the psychiatry clinic of the hospital, did not have any psychiatric disease and were in a romantic relationship.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Turkish Adaptation of Romantic Relationship Sabotage Scale (T-RSS): Validity and Reliability Study - First Evaluation | 15.01.2022-15.04.2022
  Examining the data forms and questionnaires requested from the participants between January 2022 and July 2022 and dividing the participants into three different study groups.

SECONDARY OUTCOMES:
Turkish Adaptation of Romantic Relationship Sabotage Scale (T-RSS): Validity and Reliability Study - Secondary Evaluation | 16.04.2022-15.07.2022
  Evaluating the linguistic equivalence level of the scale with the data of the first study group, performing factor analyzes and reliability studies of the scale with the data of the second and third study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Özgür MADEN, PH.D., M.D., Principal Investigator — Corresponding author
Locations (1):
- Sağlık Bilimleri Üniversitesi Sultan 2. Abdülhamid Han Eğitim ve Araştırma Hastanesi, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be sent when requested by the journal editors and reviewers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At any time
Access Criteria: After contacting the corresponding author, the data will be sent if deemed appropriate.

REFERENCES:
- [Background] Akın, A. (2012). Self-handicapping Scale: A study of Validity and Reliability. Education and Science, 37(164): 176-187.
- [Background] Arazzini Stewart, A., & De Leorge Wolker, L. (2014). Self-handicapping, perfectionism, locus of control and slef-efficacy: a path model. Pers Individ Dif, 66:160-164.
- [Background] Bowlby, J., (1973). Attachment and Loss: Separation, Anxiety and Anger. New York: Basic Books.
- [Background] Byrne, B. M. (2010). Structural Equation Modeling with Amos: Basic Concepts, Applications, and Programming (2nd ed.). New York: Taylor and Francis Group.
- [Background] Büyüköztürk, Ş. (2013). Sosyal bilimler için veri analizi el kitabı (18. baskı). Ankara: PegemA Yayıncılık.
- [Background] Büyükşahin, A., & Hovardaoğlu, S. (2004). Çiftlerin aşka ilişkin tutumlarının Lee'nin çok boyutlu aşk biçimleri kapsamında incelenmesi. Türk Psikoloji Dergisi, 19(54), 59-75.
- [Background] Conlon, E. G., Zimmer-Gembeck, M. J., Creed, P. A., & Tucker, M. (2006). Family history, self-perceptions, attitudes and cognitive abilities are associated with early adolescent reading skills. J Res Read, 29:11-32.
- [Background] Demir, M. (2008). Sweetheart, you really make me happy: Romantic relationship quality and personality as predictors of happiness among emerging adults. Journal of Happiness Studies, 9(2), 257-277. doi:10.1007/s10902-007-9051-8
- [Background] Dönmez, A.(2009). Yakın ilişkiler psikolojisi. Ankara: Nobel Yayın
- [Background] Epstein, N. B. & Baucom, D. H. (2002). Enhanced cognitive-behavioral therapy for couples: A contextual approach. Washington, DC: American Psychological Association.
- [Background] Field, A. (2009). Discovering statistics using SPSS (and sex and drugs and rock 'n' roll) (Third edition). London: SAGE Publications Ltd
- [Background] Fletcher, G. J. O., Simpson, J. A., & Thomas, G. (2000). The measurement of Perceived Relationship Quality Components: A confirmatory factor analytic approach. Personality and Social Psychology Bulletin, 26(3), 340-354. doi: 10.1177/0146167200265007
- [Background] Foster, J. J. (2001). A Beginner's Guide Data Analysis. London: Sage.
- [Background] Gottman, J. M. (1993). What predicts divorce? The relationship between marital processes and marital outcomes. Psychology Press
- [Background] Hair, J. F., Arthur H. M., Phillip, S., & Mike, P. Research Methods for Business. Chichester: John Wiley and Sons, 2007. Print.
- [Background] Hendrick, C., & Hendrick, S. (1986). A theory and method of love. Journal of Personality and Social Psychology, 50, 392-402.
- [Background] Hendrick, C., & Hendrick, S. (1990). 'A Relationship- spesific version of the Love Attitudes Scale'. Journal of Social Behavior and Personality, 5, 239-254.
- [Background] Hendrick, S., Dicke, A., & Hendrick, C. (1998). The relationships assessment scale. Journal of Social and Personal Relationships. 15(1), 137-142
- [Background] Hendrick, S. S., Hendrick, C., & Adler, N. L. (1988). Romantic Relationships: Love, Satisfaction, and Staying Together. Journal of Personality and Social Psychology, 54(6), 980-988. https://doi.org/10.1037/0022-3514.54.6.980
- [Background] Hu, L. & Bentler, P. M. (1999). Cutoff criteria for fit ındexes in covariance structure analysis: conventional criteria versus new alternatives. Structural Equation Modeling, 6(1), 1-55.
- [Background] Jones, E. E., & Rhodewalt, F. (1982). Self-Handicapping Scale [Database record]. APA PsycTests. https://doi.org/10.1037/t09528-000
- [Background] Johnson, S. M. (2004). The practice of emotionally focused couple therapy: Creating connection. (2nd ed.). New York: Brunner-Routledge.
- [Background] Karahan, A. S. (2021). Consideration of Self-Sabotage Regarding Close Relationships. OPUS International Journal of Society Researches, 18(42):1-1.
- [Background] Kearns, H., Forbes, A., Gardiner, M. L., & Marshall, K. M. (2008). When a high distinction isn't good enough: A review of perfectionism and self-handicapping. Australian Educational Researcher, 35(3):21-36.
- [Background] Kinnear, P. R. & Gray, C. D. (2006). SPSS 14 Made Simple. Oxford: Psychology Press.
- [Background] Kline, P. (2000). An easy guide to factor analysis. London and New York: Routledge.
- [Background] Lee, J. A. (1974). The styles of loving.
- [Background] Lee, J. A. (1988). Love-styles. In R.J. Sternberg, M. L. Barnes (Eds), The Psychology of Love. New Haven: Yale University Press
- [Background] Martin, K. A. & Brawley, L. R. (2002). Self-handicapping in physical achievement settings: The contributions of self-esteem and selfefficacy. Self and Identity, 1(4), 337-351. https://doi.org/10.1080/15298860290106814
- [Background] Mattingly, B. A., & Clark, E. M. (2012). Weakening relationships we try to preserve: Motivated sacrifice, attachment, and relationship quality. Journal of Applied Social Psychology, 42(2), 373-386.
- [Background] Peel, R., Caltabiano, N., Buckby, B., & McBain, K. A. (2019). Defining romantic self-sabotage: A thematic analysis of interviews with practicing psychologists. Journal of Relationship Research, 10(e16), 1-9. https://doi.org/10.1017/jrr.2019.7
- [Background] Peel, R., & Caltabiano, N. (2021a). Why do we sabotage love? a thematic analysis of lived experiences of relationship breakdown and maintenance. Journal of Couple & Relationship Therapy, 20(2), 99-131. doı: 10.1080/15332691.2020.1795039
- [Background] Sağkal, A. S., & Özdemir, Y. (2018). Turkish adaptation of perceived romantic relationshıp quality scale (prrqs): Validity and reliability study. Journal of Mehmet Akif Ersoy University Faculty of Education, (46), 22-40.
- [Background] Slade, R. (2020). Relationship Sabotage in Adults with Low Self-Esteem from Attachment Trauma in Childhood. Family Perspectives, 1(1), 11.
- [Background] Sternberg, R. J. (1986). A triangular theory of love. Psychological Review, 93(2), 119-135. https://doi.org/10.1037/0033-295X.93.2.119
- [Background] Stewart, M. A. & De George-Walker, L. (2014). Self-handicapping, perfectionism, locus of control and self-efficacy: A path model. Personality and Individual Differences, 66, 160-164. https://doi.org/10.1016/j.paid.2014.03.038
- [Background] Tabachnick, B. G., & Fidell, L. S. (2013). Using multivariate statistics (Sixth edition). United States: Pearson Education.
- [Background] Tezbaşaran, A. (1996), Likert Tipi Ölçek Geliştirme. Psikologlar Derneği Yayınları, Ankara.
- [Background] Yılmaz, B., & Gündüz, B. (2021). The differentiation of self, authenticity and depression as predictors of relationship satisfaction in emerging adulthood. Journal of Mehmet Akif Ersoy University Faculty of Education, (58), 334-361.
- [Result] Campbell L, Stanton SC. Adult attachment and trust in romantic relationships. Curr Opin Psychol. 2019 Feb;25:148-151. doi: 10.1016/j.copsyc.2018.08.004. Epub 2018 Aug 3. PMID 30096516
- [Result] Collins WA, Welsh DP, Furman W. Adolescent romantic relationships. Annu Rev Psychol. 2009;60:631-52. doi: 10.1146/annurev.psych.60.110707.163459. PMID 19035830
- [Result] Fraley RC, Hudson NW, Heffernan ME, Segal N. Are adult attachment styles categorical or dimensional? A taxometric analysis of general and relationship-specific attachment orientations. J Pers Soc Psychol. 2015 Aug;109(2):354-68. doi: 10.1037/pspp0000027. Epub 2015 Jan 5. PMID 25559192
- [Result] Peel R, Caltabiano N. The relationship sabotage scale: an evaluation of factor analyses and constructive validity. BMC Psychol. 2021 Sep 19;9(1):146. doi: 10.1186/s40359-021-00644-0. PMID 34538259